CLINICAL TRIAL: NCT06026033
Title: Does Desflurane Take Longer to Reach Target Endtidal Concentration in Patients With Higher Body Muscle Content: a Pragmatic Study
Brief Title: The Effect of Anthropometrics on Desflurane Rise Time
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Başar Erdivanlı, Assoc Prof, Recep Tayyip Erdogan University
Other Study IDs: 2022/11
Record Dates: First submitted 2023-03-31; First posted 2023-09-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Desflurane; Anesthesia, General
Keywords: Anesthetics, Inhalation; Anesthesia, General; Desflurane
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients scheduled for general anesthesia: Patients scheduled for elective general anesthesia will be included, if accepts and signs the informed consent. The inhalational anesthetic should be desflurane. No other inhalational agent should be used during the induction of anesthesia. The inspiratory and expiratory concentration of any inhalational agent should be zero before the induction of anesthesia.
  Interventions: Drug: Desflurane induction

INTERVENTIONS:
Drug: Desflurane induction — Following tracheal intubation, the fresh gas flow will be set to 1 liters/minute, desflurane vaporizer will be set to maximum.

SUMMARY:
Desflurane is increasingly used in general anesthesia. Its pharmacokinetic properties are known and its distribution is easily modeled. Yet these models fail in practice. In order to increase accuracy, any model should include cardiac output, alveolar ventilation and alveolar dead space, all of which are either hard to measure or impractical, at least.

A previous study performed by the same investigator showed that time to target endtidal concentration of sevoflurane is prolonged with increased cardiac output, but only if the patient has increased muscle mass. Although desflurane has lower muscle and fat solubility, our observations suggest a similar prolongation in case of increased muscle mass.

The investigators aim to investigate if patient characteristics such as gender, age, height, weight, body type prolongs time to reach target endtidal desflurane concentration in low flow anesthesia.

DETAILED DESCRIPTION:
Low flow anesthesia is a frequently used application in anesthesiology practice. With the widespread use of modern anesthesia devices, the implementation of this application has become easier and its complications have been greatly reduced. It is routinely applied in our clinic, accompanied by both the protocols in the literature and the protocols the investigators have created.

Desflurane is the most recently developed inhaler anesthetic agent, and it has advantages such as faster recovery from anesthesia and less metabolism compared to sevoflurane. Although the physicochemical properties of desflurane are known, computer models for its use with low-flow anesthesia are based on desflurane's physicochemical properties, and not on the pharmacokinetic properties of patients. The inhaled induction times obtained with these models do not agree with our observations in practice.

In a study conducted in 2021, it was shown that parameters such as cardiac output and alveolar ventilation can increase the accuracy of these models. Among these models, the most frequently used one in the literature is included in the Gas Man simulator, which is also used in anesthesia specialty training. It allows one to perform studies that compare simulation-based and in vivo values are carried out.

A similar study was conducted by us with sevoflurane in 2018; A significant difference was found in the rate of increase in alveolar sevoflurane concentration according to cardiac output and muscle mass. Based on this study, the investigators aimed to investigate the effect of the patient's muscle mass evaluated by pragmatic measures such as height, body weight and body type on the rate of increase in the alveolar concentration of desflurane.

For this purpose, the investigators aimed to investigate the relationship between the time to reach the targeted alveolar desflurane gas concentration and patient characteristics. The investigators believe that the results of the study will be useful in explaining the factors affecting the induction of general anesthesia with desflurane.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* planned elective surgery
* planned inhalational anesthesia
* planned use of desflurane

Exclusion Criteria:

* emergency surgery
* use of other inhalational anesthetic agent (sevoflurane, isoflurane, nitrous oxide)
* disclosed or recognized pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients, who are scheduled for elective general anesthesia. Maintenance of anesthesia with desflurane should be included in the routine anesthesia plan.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of rise in expiratory desflurane concentration | intraoperative
  Correlation between the time required for the endtidal expiratory desflurane concentration to reach 8% and patient characteristics
Rate of rise in inspiratory desflurane concentration | intraoperative
  Correlation between the time required for the endtidal inspiratory desflurane concentration to reach 6% and patient characteristics

SECONDARY OUTCOMES:
Correlation between occurrence of hypertension and patient characteristics | intraoperative
  Correlation between occurrence of hypertension defined as any measurement of systolic arterial blood pressure > 160 mmHg and patient characteristics
Correlation between occurrence of tachycardia and patient characteristics | intraoperative
  Correlation between occurrence of tachycardia defined as any measurement of heart rate > 100/minute and patient characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Başar Erdivanlı, Assoc. Prof., Study Director — Recep Tayyip Erdogan University Medical Faculty, Department of Anesthesiology and Reanimation; Alihan Madran, M.D., Principal Investigator — Recep Tayyip Erdogan University Medical Faculty, Department of Anesthesiology and Reanimation
Locations (1):
- Recep Tayyip Erdogan University Medical Faculty, Department of Anesthesiology and Reanimation, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weber J, Missbach C, Schmidt J, Wenzel C, Schumann S, Philip JH, Wirth S. Prediction of expiratory desflurane and sevoflurane concentrations in lung-healthy patients utilizing cardiac output and alveolar ventilation matched pharmacokinetic models: A comparative observational study. Medicine (Baltimore). 2021 Feb 12;100(6):e23570. doi: 10.1097/MD.0000000000023570. PMID 33578509
- [Result] Athiraman U, Ravishankar M, Jahagirdhar S. Performance of computer simulated inhalational anesthetic uptake model in comparison with real time isoflurane concentration. J Clin Monit Comput. 2016 Dec;30(6):791-796. doi: 10.1007/s10877-015-9776-6. Epub 2015 Sep 19. PMID 26386708
- [Result] Philip JH. Using screen-based simulation of inhaled anaesthetic delivery to improve patient care. Br J Anaesth. 2015 Dec;115 Suppl 2:ii89-94. doi: 10.1093/bja/aev370. PMID 26658205